CLINICAL TRIAL: NCT04492306
Title: In Vivo Clinical Evaluation of Dimethyl Sulfoxide Dentin Pre-treatment Prior to a Two-step Etch and Rinse Adhesive: Randomized Controlled Trial
Brief Title: Clinical Evaluation of Dimethyl Sulfoxide Dentin Pre-treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: University of Turku (Other)
Responsible Party: Principal Investigator, Omar Abdelaziz Ismail, Assistant Lecturer of Restorative Dentistry,HUE. Member of the adhesive group of Turku., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMSO Clinical Trial
Record Dates: First submitted 2020-07-22; First posted 2020-07-30 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Dental Diseases
Keywords: DMSO
MeSH Terms: conditions — Stomatognathic Diseases | interventions — Dimethyl Sulfoxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: In our clinical trial double blinding will be performed, the participants and both assessors (H.M.& N.H.) will be blinded to the type of the material used to reduce performance and ascertainment bias and also reduce biased estimates of treatment effects. The operator cannot be blinded in this trial because of the difference in the application procedures of each restorative material. Therefore, the operator (O.I.) will take care to treat the two allocation groups as equally as possible by standardizing the care of participants, frequency of follow-ups and management of complications.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3M single bond, etch and rinse adhesive (Active Comparator): O.I. will clean the labial surface of tooth with polishing paste and brush Roughening of the surface may be needed by diamond point The tooth will be isolated by rubber dam. Apply etchant for 30 s for enamel and 15 s for dentin. Rinse thoroughly with water for 10 s. blot-drying with paper tissue was carefully performed leaving the dentin surface slightly moist.
  Apply 2 to 3 consecutive coats of the adhesive for 15 s. Gently air for 5 s. Light cure for 10 s. Composite build ups (Filtek Z350 XT, 3 M ESPE, St Paul, MN, USA) were performed in increments and individually light-cured for 40 s. Light curing of all resin materials was performed using a LED device (Bluephase 20i, Ivoclare Vivadent, Schaan, Liechtenstein) delivering 1100 mW/cm2.
  Interventions: Other: 3M ESPE Single bond 2; Other: Filtek Z350 XT, 3 M ESPE, St Paul, MN, USA); Other: 3m ESPE etch
- DMSO pre-treatment before 3M single bond application (Experimental): The same steps of the comparator group with additional step, after dentin etching and humidity control, dentin pretreatments were performed consisting of active application of 1% DMSO/H2O solutions on etched-dentin followed by blot drying until paper filters no longer absorbed liquids from the bonding surface by capillarity then apply adhesive.
  Interventions: Other: Dimethyl Sulfoxide; Other: 3M ESPE Single bond 2; Other: Filtek Z350 XT, 3 M ESPE, St Paul, MN, USA); Other: 3m ESPE etch

INTERVENTIONS:
Other: Dimethyl Sulfoxide — DMSO [(CH3)2SO] is a polar aprotic solvent that dissolves both polar and non-polar compounds.
  Other Names: 1% DMSO
  Arms: DMSO pre-treatment before 3M single bond application
Other: 3M ESPE Single bond 2 — Total etch adhesive bond
Other: Filtek Z350 XT, 3 M ESPE, St Paul, MN, USA) — Composite Resin
Other: 3m ESPE etch — 32% phosphoric acid

SUMMARY:
This study is conducted in order to evaluate the clinical effectiveness of 1% DMSO dentin pre-treatment on the clinical performance of etch and rinse adhesive.

DETAILED DESCRIPTION:
Despite substantial advances in resin-dentin bonding over the past decades, reduction in bonding effectiveness of currently available dental adhesives remains a major limitation in modern adhesive dentistry. Hydrolysis of both organic and resin constituents of hybrid layer persists as impediments in dentin bonding longevity. Since bonding is directly related to the quality of the formed polymer the resin components play an important role in proper resin-dentin interaction and in the mechanical properties of the material.

In face of the limitations of most current clinically-feasible bonding protocols and inherent drawbacks of the etch-and-rinse approach an ideal resin-enveloped collagen scaffold is unlikely to be produced in a consistent manner. In dentin hybridization, adhesive infiltration is far from perfect resulting in poorly formed hybrid layers. Replacement of all 70 vol% residual water in etched-dentin with monomers is hardly achieved. For this reason, the hybrid layer may be considered as the weak link in resin-dentin bonds.

DMSO [(CH3)2SO] is a polar aprotic solvent that dissolves both polar and non-polar compounds. It is a polyfunctional molecule, with a highly polar S O group and two hydrophobic methyl groups, fully miscible in most solvents and monomers used in adhesive dentistry. DMSO is perhaps the best currently known penetration enhancer for medical purposes with the ability to dissociate the highly crosslinked collagen into a sparser network of apparent fibrils.

The rationale for testing a bonding resin with relatively low DMSO-content is that incorporation of high DMSO concentrations may hamper the mechanical properties of dimethacrylate bonding polymers, which in turn could compromise the bonded interface. DMSO's ability to "biomodify" collagen structure, increasing spaces between collagen microfibrils and improving dentin wettability support the improved bonding effectiveness even under dry-conditions. It is evident that this simplified use of DMSO or, to a better extent, its use as a dentin pretreatment reduced technique sensitivity of the etch-and-rinse approach concomitantly allowing water removal from the bonded interface by the proposed dry-bonding technique. Optimized bonding efficiency combined with reduced water-content during dentin hybridization could greatly contribute to clinical long-term durability.

Nevertheless, further studies are necessary to test such hypothesis. Specially that there is no clinical study support this theory yet even DMSO had taken the FDA approval many years ago as a pharmaceutical solvent and has been used in several medications. DMSO caused no or minor cytotoxic effects on the pulp tissue repair-related activity of odontoblast-like cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cervical lesions.
* Co-operative patients approving to participate in the study.
* Pulp is asymptomatic vital teeth.
* Presence of favorable occlusion and teeth are in normal contact with the adjacent teeth.

Exclusion Criteria:

* Xerostomia.
* Bruxism and visible wear facets in the posterior dentition.
* Known inability to return for recall appointments.
* Fractured or visibly cracked candidate tooth.
* Current desensitizing therapy, including desensitizing dentifrices or other over-the-counter (OTC) products.
* Long-term use of anti-inflammatory, analgesic, or psychotropic drugs.
* Pregnancy or breastfeeding (potential conflicts with recall dates.
* Allergies to ingredients of resin-based restorative materials.
* Orthodontic appliance treatment within the previous three months.
* Abutment teeth for fixed or removable prostheses.
* Teeth or supporting structures with any symptomatic pathology.
* Existing periodontal disease or periodontal surgery within the previous three months.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Biological (change of caries adjacent to the restoration) | Day 0, Month 6, Month 12, Month 18
  FDI criteria for evaluation of restorations, percentage score.
  * Score: Properties
  * Clinically excellent/ very good: No secondary or primary caries.
  * Clinically good: Small and Localized 1. Demineralization, 2. Erosion or 3. Abfraction.
  * Clinically sufficient/satisfactory: Larger areas Of 1. Demineralization, 2. Erosion or 3. Abrasion/abfraction, dentine not exposed.
  * Clinically unsatisfactory: Caries with Cavitation and suspected undermining caries, 2. Erosion in dentine, 3. Abrasion/ abfraction in dentine.
  * Clinically poor: Deep caries or exposed dentine that is not accessible for repair of restoration.

SECONDARY OUTCOMES:
Functional (change of marginal adaptation) | Day 0, Month 6, Month 12, Month 18
  FDI criteria for evaluation of restorations, percentage score.
  * Score: Properties.
  * Clinically excellent/ very good: Harmonious outline, no gaps, no white or discolored lines.
  * Clinically good: Marginal gap (<150 µm), White lines. Or Small marginal fracture removable by polishing. or Slight ditching, slight step/flashes, minor Irregularities.
  * Clinically sufficient/satisf actory: Gap < 250 µm not removable. Or Several small marginal fractures. Or Major irregularities, ditching or flash, steps.
  * Clinically unsatisfactory: Gap > 250 µm or dentine/base exposed. Or Severe ditching or marginal fractures. or Larger irregularities or steps (repair necessary).
  * Clinically poor: Restoration (complete or partial) is loose but in situ. Or Generalized major gaps or irregularities.

OTHER OUTCOMES:
Esthetic (Color match and translucency) | Day 0, Month 6, Month 12, Month 18
  FDI criteria for evaluation of restorations, percentage score.
  * Score: Properties
  * Clinically excellent/ very good: Good color match, no difference in shade and/or translucency.
  * Clinically good: Minor deviations in shade and/or translucency.
  * Clinically sufficient/satisfactory: Distinct deviation but acceptable. Does not affect esthetics: 1. more opaque ,2. more translucent ,3. darker,4. brighter.
  * Clinically unsatisfactory: Localized clinically deviation that can be corrected by repair: 1.Too opaque, 2.Too translucent,3. Too dark, 4.Too bright.
  * Clinically poor: Unacceptable. Replacement necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Randa Hafez, Professor, Study Director — Cairo U
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt